CLINICAL TRIAL: NCT04066192
Title: A Pharmacogenetic Human Laboratory Investigation of Brexpiprazole in Alcohol Use Disorder
Brief Title: Brexpiprazole in Alcohol Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-1658; 1R01AA027765-01 (NIH)
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — brexpiprazole

STUDY DESIGN:
Intervention Model Description: Double-blind placebo controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be blind to medication assignment, as will all care providers and investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Participants in this Arm will take a medically inert placebo. To ensure pill equivalence between groups, tablets will be packaged in the same capsule; thus, each participant will take one capsule per day. Participants will be instructed to ingest the capsule orally each morning.
  Interventions: Drug: Placebo
- BREX 2mg (Active Comparator): The BREX 2mg group will start at the same dose at the BREX 4mg group and titrate up at the same rate, so the BREX 2mg Arm will take .5 mg of brexpiprazole on day 1-2, 1 mg on day 3-4, and 2mg on day 5, to reach its final 2mg dose for day 5-14. To ensure pill equivalence between groups, tablets will be packaged in the same capsule; thus, each participant will take one capsule per day. Participants will be instructed to ingest the medication orally each morning.
  Interventions: Drug: Brexpiprazole
- BREX 4mg (Active Comparator): The BREX 4mg group will start at the same dose as the BREX 2mg group and titrate up at the same rate, so the BREX 4mg Arm will take .5 mg of brexpiprazole on day 1-2, 1 mg on day 3-4, 2mg on day 5-6, and 4mg on day 7 to reach its final 4mg dose for days 7-14. To ensure pill equivalence between groups, tablets will be packaged in the same capsule; thus, each participant will take one capsule per day. Participants will be instructed to ingest the medication orally each morning.
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole will be used in .5mg, 1mg, 2mg, and 4mg doses as described in the study arms.
  Arms: BREX 2mg; BREX 4mg
Drug: Placebo — A medically inert placebo medication will be used as described in the study arms.
  Arms: Placebo

SUMMARY:
Few medications are currently Food & Drug Administration (FDA)-approved for the treatment of Alcohol Use Disorder (AUD), and those that are have, on average, modest effects on drinking. "Precision medicine" research has explored whether patient-level variables, such as genetic variation, may identify subgroups of individuals with larger medication effects, but few findings have been replicated. A promising novel medication for AUD is brexpiprazole (BREX), a serotonin/dopamine activity modulator (SDAM). The investigators conducted a prior study in which the effects of another SDAM, aripiprazole, were influenced by genetic variation in the gene encoding the dopamine transporter (DAT1). This study will evaluate the effects of two doses of BREX, relative to placebo, among non-treatment-seeking individuals with AUD, and will test whether DAT1 genotype influences these effects. Primary outcomes are drinking under natural conditions and in a laboratory paradigm. Functional magnetic resonance imaging (fMRI) will be used to explore whether BREX effects on brain activation associated with cognitive control or elicited by alcohol cues accounts for its effects on drinking. The investigators hypothesize that BREX, relative to placebo, will reduce drinking under natural conditions and in the lab, and will do so to a greater extent among individuals who carry the DAT1 9-repeat allele, relative to those homozygous for the 10-repeat allele. If these hypotheses are supported, BREX may represent a novel pharmacogenetic treatment for AUD.

DETAILED DESCRIPTION:
The overarching hypothesis of this study is that brexpiprazole (BREX) (2 or 4 mg/day), relative to placebo, will reduce alcohol consumption and modulate the neural substrates of moderate-severe Alcohol Use Disorder (AUD), and that genotype at a variable number tandem repeat polymorphism (VNTR) in the DAT1/SLC6A3 gene will predict BREX effects. Participants will be non-treatment-seeking AUD individuals, and will be prospectively randomized to medication on the basis of their DAT1 VNTR genotype. Since BREX affects both cortical and striatal neurophysiology, the investigators will use functional magnetic resonance imaging (fMRI) to test its effects on cortical (right inferior frontal gyrus; rIFG) activation associated with response inhibition and on striatal activation elicited by alcohol cues, and will explore whether either of these measures mediates BREX effects on drinking in the natural environment vs. a bar-lab setting, which may reflect different aspects of lost control over drinking.

Aim 1: Test BREX effects on inhibition-related cortical activation and alcohol cue-elicited striatal activation, and evaluate whether DAT1 VNTR genotype predicts these effects.

Hypothesis 1: There will be a linear effect of BREX dose, relative to placebo, in increasing inhibition-related rIFG activation and reducing cue-elicited ventral striatum (VS) activation, and these effects will be greater among DAT1 9R carriers than 10R homozygotes.

Aim 2: Test BREX effects on drinking in the natural environment and alcohol self-administration in the bar lab, and evaluate whether DAT1 VNTR genotype predicts these effects.

Hypothesis 2: There will be a linear effect of BREX dose, relative to placebo, in reducing natural drinking and alcohol self-administration, and these effects will be greater among DAT1 9R carriers.

Aim 3: Test inhibition-related cortical activation and cue-elicited VS activation as mechanisms of action for BREX's effects on natural and bar-lab drinking.

Hypothesis 3: Cue-elicited VS activation will mediate BREX effects on natural drinking, while inhibition-related rIFG activation will mediate its effects on bar-lab drinking.

This study will recruit up to 250 study participants with Alcohol Use Disorder (AUD) who are not seeking treatment for AUD. Individuals will complete an initial phone screen to assess inclusion/exclusion criteria that can be determined over the phone, and eligible participants will subsequently be scheduled for an in-person screening session. After giving informed consent, participants will complete a medical screening and psychiatric assessment, and biological samples (blood and urine) will be collected. Participants who remain eligible after this screening session will be randomly assigned to take one of two doses of brexpiprazole (2 milligram (mg) or 4 mg per day) or matched placebo for 14 days. Both investigators and participants will be blind to medication group assignments. After the in-person screening session, there are five study visits. 1) Day 1 of study medication: participants will complete a one-hour-long functional magnetic resonance imaging (fMRI) brain scan and take the first dose of study medication. 2) Day 7: participants will return to the lab for a brief check-in at which medication side effects will be assessed. 3) Day 13: blood and urine samples will be collected again; participants will take that day's dose of medication in the lab and then complete another one-hour-long fMRI brain scan. 4) Day 14: participants will take the last dose of medication in the lab and then complete a day-long procedure in which alcohol will be administered. 5) Day 15: participants will be debriefed and compensated $600 for study participation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-65.
* Meet DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th edition) diagnostic criteria for AUD, as assessed by the Structured Clinical Interview for DSM-5 (SCID-5).
* Currently not engaged in, and does not want treatment for, AUD.
* Currently not taking any medication for AUD.
* Able to read and understand questionnaires and informed consent.
* Lives within 50 miles of the study site.
* Physically healthy with no history of significant medical illness.
* Negative urine drug screen (UDS) for all substances of abuse prior to taking the first dose of medication.

Please contact clinical site for additional inclusion criteria.

Exclusion Criteria:

* Refusal of valid written consent.
* Insufficient English skills for consenting or interviews.
* Severe claustrophobia or morbid obesity that preclude placement in the MRI scanner.
* Contraindications to MRI scanning, ferrous metal in the body including intracranial, intraorbital, or intraspinal metal, pacemakers, cochlear implants or other non-MRI-compatible devices.
* History of head injury with loss of consciousness for more than 2 minutes, neurological illness, or history of neurosurgical procedures.
* Current DSM-5 diagnosis of any other substance use disorder except Nicotine Use Disorder.
* Current DSM-5 psychotic, mood, anxiety, obsessive-compulsive, trauma-related, or eating disorder, as assessed by SCID-5.
* Current suicidal ideation or homicidal ideation.
* Current use of any psychoactive medication, as evidenced by self-report and UDS.
* History of severe alcohol withdrawal (e.g., seizure, delirium tremens), as evidenced by self-report and assessment with Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar).
* Clinically significant medical problems such as cardiovascular, renal, gastrointestinal, or endocrine problems, as evidenced by medical history and physical exam.
* Past alcohol-related medical illness, such as gastrointestinal bleeding, pancreatitis, or peptic ulcer.
* Current or past hepatocellular disease, as indicated by verbal report or elevations of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 3 times the upper limit of the normal range at screening.
* Females of childbearing potential who are pregnant (by plasma or urine HCG), nursing, or who are not using a reliable form of contraception.
* Current charges pending for a violent crime (not including DUI-related offenses).
* Currently incarcerated.
* Lack of a stable living situation.
* History of head injury with loss of consciousness for more than 2 minutes, neurological illness, or history of neurosurgical procedures.
* Decisionally challenged.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of drinks consumed in natural environment | First 13 days of medication period
  The number of standard alcoholic drinks participants consume during the first 13 days of the medication period, as reported on the Timeline Follow-Back Interview.
Number of drinks consumed in bar lab | Day 14 of medication period
  The number of drinks (out of 8 possible) that participants choose to consume in the bar lab.
Change in alcohol cue-elicited brain activation (fMRI) | 14 days - change between baseline and day 14 scan.
  Magnitude of change between baseline and day 14 fMRI scan in the blood oxygenation level dependent (BOLD) signal to alcohol cues, relative to neutral beverage cues on the Alcohol Cue Reactivity Task.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Schacht, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, individual-level phenotypic data will be submitted to the NIAAA Data Archive (NDA) portal once it is available, and genotypic data (e.g., DAT1 genotypes and any other genomic data generated from study participants' whole blood samples) will be submitted to the NIH dbGAP repository. Informed consent that allows for broad sharing of each subject's de-identified data will be obtained and personally identifiable information that allows the creation of an NDA Global Unique Identifier will be collected. Study staff will work with NDA staff to specify and/or define measures to be collected (including the manner in which raw and pre-processed neuroimaging data will be shared), and data will be submitted in accordance with NDA submission due dates.
Time Frame: Data will become available 2 years after the grant end date, and will be available as long as the NDA exists.
Access Criteria: Investigators at institutions with a Federal Wide Assurance (FWA) will be able to gain access to NDA data by submitting a data access request in accordance with applicable NDA policies (see https://ndar.nih.gov/access.html for sample policies). Data requests will be reviewed and granted by a NIAAA Data Access Committee.

REFERENCES:
- [Background] Schacht JP, Voronin KE, Randall PK, Anton RF. Dopaminergic Genetic Variation Influences Aripiprazole Effects on Alcohol Self-Administration and the Neural Response to Alcohol Cues in a Randomized Trial. Neuropsychopharmacology. 2018 May;43(6):1247-1256. doi: 10.1038/npp.2017.298. Epub 2017 Dec 6. PMID 29362512